CLINICAL TRIAL: NCT02561572
Title: The Effect of Acupuncture on Pre-operative Anxiety Levels in Neurosurgical Patients: a Randomised, Controlled Trail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STH19048
Record Dates: First submitted 2015-09-25; First posted 2015-09-28 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-02

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Acupuncture at the Yintang point for 30 minutes.
  Interventions: Other: Acupuncture
- Control (No Intervention): No intervention for 30 minutes.

INTERVENTIONS:
Other: Acupuncture — Yintang point acupuncture
  Arms: Intervention

SUMMARY:
Preoperative anxiety has been associated with adverse consequences, including increased anaesthetic and analgesic requirements and overall dissatisfaction with care. Traditionally this has been treated with sedative drugs, such as benzodiazepines, but these can be associated with a sedative "hangover" with sedation continuing into the postoperative period. This is undesirable in patients undergoing neurosurgical procedures, as there is a need to assess neurological status in the immediate postoperative period. Acupuncture at the Yintang point (on the forehead between the eyebrows) has been shown to effectively reduce preoperative anxiety, but studies undertaken in the United Kingdom and neurosurgical population are lacking. The investigators aim to investigate the effect of acupuncture at the Yintang point on preoperative anxiety. Anxiety levels will be measured using two validated questionnaires: the State-Trait Anxiety Inventory (STAI) and Amsterdam Preoperative Anxiety and Information Scale (APAIS).

DETAILED DESCRIPTION:
1. Methodology All patients presenting for neurosurgery will be considered and the study will take place on the Theatre Admissions Units at the Royal Hallamshire Hospital, Sheffield, United Kingdom. After gaining consent, baseline anxiety levels will be assessed using the APAIS and STAI questionnaires. The subject will then be randomised using a web-based programme to one of two groups: intervention (Yintang point), or control (no intervention). All the acupuncture will done with the same type of needle and by the same investigator. The questionnaires will be repeated 30 minutes later to assess the effect of the intervention.
2. Design: type of study design and justification The study is a randomised control trial looking at an acupuncture point utilised for anxiety reduction (Yintang), and a controls. The ratio of intervention to controls is 1:1. After advice for experts in acupuncture, the investigators are not including a placebo acupuncture intervention or sham acupuncture. This is because it is increasingly recognised that any form of acupuncture or acupressure can have central effects and that sham acupuncture is actually impossible to undertake. Pilot study data (awaiting publication) done in the investigator's institution demonstrated a mean (standard deviation) STAI score in neurosurgical patients of 8.86 (4.4). Previous data have suggested that acupuncture may reduce anxiety levels by 25-37%. Assuming a p< 0.05 and power 0.9, in order to demonstrate a 30% reduction in STAI scores, the investigators will need 58 patients in each group. Assuming a 10% dropout rate, the investigators aim to recruit 64 patients in each group (128 in total). The investigators have shown that anxiety levels are not related to gender or site of surgery (cranial vs. spinal) and therefore will not stratify the groups. The investigators will undertake block randomisation to try and minimise any learning effects by the acupuncturist.
3. Analysis including statistical methods, where appropriate The investigators will use analysis of variance (ANOVA) to analyse anxiety scores from the two questionnaires (after testing for normality of data distribution). Pain scores will be analysed by t-tests and postoperative nausea and vomiting (PONV) incidence by Chi-squared.

ELIGIBILITY:
Inclusion Criteria:

- Undergoing neurosurgical procedure under general anaesthesia

Exclusion Criteria:

* pregnancy
* psychiatric disorders
* inability to provide own consent
* the use of sedative medication (benzodiazepines or sleeping tablets) in the 24 hours prior to surgery
* previous acupuncture experience
* any contraindication to the use of acupuncture such as bleeding disorders or skin inflammation/infection at the treatment sites
* use of preoperative acupuncture for other reasons (prevention of postoperative nausea and vomiting).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Wiles, BM BS FRCA, Study Chair — Consutant, Sheffield Teachinh Hospital NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospital NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 64 | 64
Completed | 62 | 62
Not Completed | 2 | 2
Not completed — Inadequate time before surgery | 2 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (13.6) | 54 (17.5) | 54.7 (15.7)
Sex/Gender, Customized [Number; unit: participants]
  Female | 36 | 32 | 68
  Male | 26 | 30 | 56

OUTCOME MEASURES:

1. Primary Outcome: State-Trait Anxiety Inventory Score
Description: Patients completed the six item short form of the State-Trait Anxiety Inventory (STAI-S6) in order to assess baseline anxiety levels prior to any intervention. The STAI-S6 is a standardised short form of the 40-item Spielberger State-Trait Anxiety Inventory that has three anxiety-present and three anxiety-absent questions (Table 1). Scores from the STAI-S6 are prorated up to allow comparison with the full version of the questionnaire, with scores ranging from 20 (low anxiety) to 80 (high anxiety). The STAI-S6 has been shown to correlate well with the full version, [12] but is much quicker for participants to complete.
Time Frame: 30 minutes after intervention
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 62 | 62
units on a scale | 40.0 [30.0 to 46.7] | 43.3 [36.7 to 50.0]

2. Secondary Outcome: Amsterdam Preoperative Anxiety and Information Scale Scores
Description: The Amsterdam Pre-operative Anxiety and Information Scale has four questions relating to anxiety (APAISa, Table 2) and has been shown to correlate well with the full version of the State-Trait Anxiety Inventory. The scores from the anxiety elements of the questionnaire are added together giving a possible of total score of 4 (low anxiety) to 20 (high anxiety).
Time Frame: 30 minutes after intervention
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 62 | 62
units on a scale | 7 [4 to 10] | 8.5 [6 to 12]

3. Secondary Outcome: Incidence of Postoperative Nausea and Vomiting (PONV) in the Postanaesthetic Care Unit (PACU)
Time Frame: Within 30 minutes of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 57 | 49
Participants | 2 | 1

4. Secondary Outcome: Incidence of Postoperative Nausea and Vomiting (PONV)
Time Frame: 24 h postop
Population: Unable to collect data on wards after discharge from PACU
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Pain Score in the Postanaesthetic Care Unit (PACU)
Description: The number of patients experiencing moderate/severe pain in PACU.
Time Frame: Immediately postop
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 57 | 49
Participants | 28 | 21

6. Secondary Outcome: Pain Score
Time Frame: 24 h postop
Population: Unable to collect data on wards after PACU discharge.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 0/62 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes